CLINICAL TRIAL: NCT03387371
Title: Clinical and Microbiologic Effects of Nonsurgical Periodontal Treatment Combined With an Erbium: Yttrium Aluminium Garnet Laser
Brief Title: Laser Assisted Nonsurgical Periodontal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LaserPerio001
Record Dates: First submitted 2017-11-07; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-11

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis, laser
MeSH Terms: conditions — Chronic Periodontitis | interventions — Ultrasonography; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasonics & Gracey Curettes (Active Comparator): Scaling and root planning is done with ultrasonics and gracey curettes in 24 hours with two visits.
  Interventions: Device: Ultrasonics; Device: Gracey Curettes
- Ultrasonics & Gracey Curettes & Laser (Experimental): Scaling and root planning is done with ultrasonics, gracey curettes and Er:YAG laser in 24 hours with two visits.
  Interventions: Device: Gracey Curettes; Device: Er:YAG Laser

INTERVENTIONS:
Device: Ultrasonics — ultrasonic scalers
  Arms: Ultrasonics & Gracey Curettes
Device: Gracey Curettes — Spesific gracey curettes
Device: Er:YAG Laser — 2940 nm wavelenght Er:YAG laser
  Arms: Ultrasonics & Gracey Curettes & Laser

SUMMARY:
Periodontitis is a chronic inflammatory disease caused by mixed infections with the subgingival microbiota being organized as a biofilm that, if untreated, may result in breakdown of the periodontal tissues in susceptible individuals. Evidence from intervention studies shows that mechanical root debridement significantly improves periodontal health by halting the progression of periodontal tissue breakdown. In order to improve effectiveness and efficacy of the removal of the subgingival biofilm, Er:YAG laser therapy has recently been recommended as an alternative to conventional scaling procedures.

ELIGIBILITY:
Inclusion Criteria:

Greater than 25 years, Clinical diagnosis of moderate to advanced chronic periodontitis, Pocket depth ≥ 5 mm or clinic attachment level ≥ 4 mm at least in two interproximal areas (not on the same tooth), Along with very good oral hygiene scores (GI≤1and PI≤1), At least 4 teeth in each quadrant, Teeth with subgingival plaque sample is collected has no restoration or prothesis

Exclusion Criteria:

Periodontal treatment ( root planning or surgical periodontal treatment) had done before, Systemic disease that could influence the outcome of periodontal therapy, Prophylaxis regime mandatory during periodontal treatment, Use of any drug that could influence the outcome of periodontal therapy, Use of antibiotics within the last 3 months, Use of anti-inflammatory drugs within the last 3 months, Use of removable prothesis Pregnancy, lactation or use of hormone contraceptives, Smoking

Ages: 28 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-01-20 (Estimated); Study Completion 2018-01-20 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth 3 | 3. month
  to measure the probing pocket depth of all teeth
Clinic Attachment Level 3 | 3. month
  to measure the Clinic Attachment Level of all teeth
Subgingival Plak Sample 1 | 1. month
  quantitative changes on red complex bacterias
Probing Pocket Depth 6 | 6. month
  to measure theProbing Pocket Depth of all teeth
Clinic Attachment Level 6 | 6. month
  to measure the Clinic Attachment Level of all teeth
Subgingival Plak Sample 3 | 3. month
  quantitative changes on red complex bacterias
Subgingival Plak Sample 6 | 6. month
  quantitative changes on red complex bacterias

SECONDARY OUTCOMES:
Bleeding On Probing 3 | 3. month
  to record the Bleeding On Probing of all teeth
Bleeding On Probing 6 | 6. month
  to record the Bleeding On Probing of all teeth
Plak Index 3 | 3. month
  to record the plak index of all teeth
Plak Index 6 | 6. month
  to record the plak index of all teeth

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zengin Celik T, Saglam E, Ercan C, Akbas F, Nazaroglu K, Tunali M. Clinical and Microbiological Effects of the Use of Erbium: Yttrium-Aluminum-Garnet Laser on Chronic Periodontitis in Addition to Nonsurgical Periodontal Treatment: A Randomized Clinical Trial-6 Months Follow-Up. Photobiomodul Photomed Laser Surg. 2019 Mar;37(3):182-190. doi: 10.1089/photob.2018.4510. Epub 2019 Feb 21. PMID 31050949